CLINICAL TRIAL: NCT01425944
Title: The Brain Vascular Malformations Clinical Research Network: Predictors of Clinical Course, Project 2: Innovative Approaches to Gauge Progression of Sturge-Weber Syndrome
Brief Title: Innovative Approaches to Gauge Progression of Sturge-Weber Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California, San Francisco (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Duke University (Other); Children's Hospital of Michigan (Other); Baylor College of Medicine (Other); Wills Eye (Other); Nationwide Children's Hospital (Other); New York University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Anne Comi, MD, Principal Investigator, Director Sturge-Weber Center, Kennedy Krieger Institute, Professor Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Other Study IDs: NA_00038014; U54NS065705-02 (NIH); BVMC6202 (Other: Rare Diseases Clinical Research Network); BVMC6208 (Other: Rare Diseases Clinical Research Network)
Record Dates: First submitted 2011-08-29; First posted 2011-08-30 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2024-02

CONDITIONS: Sturge-Weber Syndrome
Keywords: Sturge Weber Syndrome; Biomarkers; DNA arrays; brain vessel malformations
MeSH Terms: conditions — Sturge-Weber Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Aim 1 retains data and samples without DNA. Aim 2 retains data without DNA. Aim 3 retains anonymous data with DNA.
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
This study has three aims that hope to expand the knowledge on the cause of Sturge-Weber Syndrome (SWS) and improve clinical care of Sturge-Weber Syndrome patients.

DETAILED DESCRIPTION:
This study is one of three projects of an NIH Rare Disease Clinical Research Consortium focused on brain blood vessel malformations in three different rare diseases. The focus of this project is on Sturge-Weber Syndrome.

We plan to improve the future understanding and treatment of Sturge-Weber Syndrome by 1) establishing a national consortium database which will gather lager amounts of clinical data and serve indirectly as a registry to foster future clinical trials and determine the usefulness of urine vascular biomarkers to determine the vascular remodeling of the SWS birthmark and choroidal angioma, 2) study vascular remodeling with retrospective and prospective neuroimaging to determine the vascular remodeling of the deep draining intraparenchymal vessels as it relates to SWS neurologic status, and 3) relate the GNAQ mutation to altered phosphorylation of pathway proteins and angiogenesis factors in SWS tissue.

ELIGIBILITY:
Inclusion Criteria:

For Aim 1:

For main sample:

* Sturge-Weber syndrome
* Diagnosed brain Involvement

For Control:

* Family member of participating SWS patient

For OCT:

* Sturge-Weber syndrome eye involvement

For Aim 2:

* Sturge-Weber syndrome
* Diagnosed Brain Involvement

For Aim 3:

* Sturge-Weber syndrome
* Diagnosed brain Involvement
* Port-Wine Stain in V1 and/or V2 areas of face.

Exclusion Criteria:

* Not Diagnosed with Sturge-Weber syndrome with brain Involvement (or eye involvement for OCT)

For Aim 1:

* Family member must not have certain medical conditions. A list will be provided before consent is given.

For Aim 3:

* Not Diagnosed with Sturge-Weber syndrome with brain Involvement
* No Port-Wine Stain

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For Aim 1, the population will be subjects with Sturge-Weber Syndrome and diagnosed brain involvement. There will be a separate group made up of family members of those with Sturge-Weber syndrome brain involvement to have as a control for the urine portion of Aim 1. For the optical coherence tomography (OCT) portion of Aim 1, the population will be subjects with Sturge-Weber Syndrome eye involvement. For Aim 2, the population will be subjects that have Sturge-Weber Syndrome with brain involvement. For Aim 3, the population will be subjects with Sturge-Weber Syndrome, diagnosed brain involvement, and V1 distribution Port-Wine Stain.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Aim 1 | All 5 years
  Descriptive statistics for the national database, correlation between neurologic score and urine angiogenesis factor, and correlation between PWS (port-wine stain) attributes, urine vascular factors, and neuroscore
Aim 2 | All 5 years
  Correlation between neuroscore and degree of collateral venous vessel opening
Aim 3 | All 5 years
  Correlation between GNAQ mutation status and hyperphosphorylation in downstream proteins

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Comi, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (7):
- United States (7):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Wayne State University/Children's Hospital of Michigan, Detroit, Michigan
  - New York University, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Wills Eye Institute, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No